CLINICAL TRIAL: NCT03676712
Title: The Effect of Flexible Thoracolumbar Brace on Idiopathic Scoliosis, Prospective, Randomized, Open-label Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of subjects was not successful.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: B-1805/471-002
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- scoliosis patients (Experimental): scoliosis patients who have cobb angle over 20 degree wear scoliosis brace for six months
  Interventions: Device: scoliosis brace

INTERVENTIONS:
Device: scoliosis brace — Wear at least 18 hours a day

SUMMARY:
The Effect of Flexible Thoracolumbar Brace on Idiopathic Scoliosis, Prospective, Randomized, Open-label Trial

ELIGIBILITY:
Inclusion Criteria:

* who have idiopathic scoliosis, showing at Cobb's angle over 20 degrees,less than 45 on X-ray

Exclusion Criteria:

* Patients who underwent spinal surgery
* Patients with spinal scoliosis due to cerebral palsy, muscle paralysis, polio, congenital spinal abnormalities
* Patients observed with Cobb's angle less than 20 degrees, over 45 degrees
* Patients complaining of acute low back pain
* Patients with cognitive impairment, severe mental illness, and inability to communicate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
cobb angle | through study completion, an average of 6 months
  measure lateral curve of vertebra on spine x-ray AP view

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea